CLINICAL TRIAL: NCT03995706
Title: A Phase 0, Investigator Initiated Study to Determine the Bioavailability of Sacituzumab Govitecan in Breast Brain Metastasis and Glioblastoma
Brief Title: Neuro/Sacituzumab Govitecan/Breast Brain Metastasis/Glioblastoma/Ph 0
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 19-0069; HSC20190378H (Other: UT Health Science Center Institutional Review Board)
Record Dates: First submitted 2019-06-17; First posted 2019-06-24 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Breast Brain Metastasis and Glioblastoma (Experimental): Sacituzumab Govitecan treatment will be initiated with a 10mg/kg standard dose without any dose escalation on day-1, prior to surgery. Sacituzumab govitecan and will continue to be administered by IV infusion over 3 hours on Days 1 and 8 of a 21 day cycle post-operatively until progression.
  Interventions: Drug: Sacituzumab Govitecan

INTERVENTIONS:
Drug: Sacituzumab Govitecan — All 20 subjects will receive study drug Sacituzumab Govitecan preoperatively. Intraoperative tissue collection will follow with contemporaneous CSF (depending on tumor location) and whole blood (serum) sampling. Samples will be tested for total SN-38and free SN-38, as well as SN-38G. Following recovery from surgery, patients will resume treatment

SUMMARY:
Single center, non-randomized, Phase 0 study. Sacituzumab Govitecan given preoperatively, followed by craniotomy with surgery or biopsy of brain tumors (GBM and metastatic brain tumors from Breast) and intraoperative tissue collection will follow with contemporaneous CSF (depending on tumor location) and whole blood (serum) sampling.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Histologically or cytologically documented breast cancer (Cohort A) with known or suspected parenchymal brain metastases.
* Recurrent glioblastoma (Cohort B) with documented progression by RANO criteria following standard combined modality treatment with radiation and temozolomide.
* Plans to undergo craniotomy as part of standard of care. Patients emergently needing surgical debulking due to symptoms of their disease are not eligible.
* Recovered from toxicities of prior therapy to grade 0 or 1
* ECOG performance status ≤ 2.
* Life expectancy of at least 3 months.
* Acceptable liver function:
* Bilirubin ≤ 1.5 times upper limit of normal
* AST (SGOT) and ALT (SGPT) ≤ 3.0 times upper limit of normal (ULN);
* Adequate renal function: calculated creatinine clearance ≥30mL/minute according to the Cockcroft and Gault formula
* Acceptable hematologic status (without hematologic support)
* ANC ≥1500 cells/uL
* Platelet count ≥100,000/uL
* Hemoglobin ≥9.0 g/dL
* All women of childbearing potential must have a negative serum pregnancy test and male and female subjects must agree to use effective means of contraception (surgical sterilization or the use or barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose.

Exclusion Criteria:

* The subject is receiving warfarin (or other coumarin derivatives) and is unable to switch to low molecular weight heparin (LMWH) before the first dose of study drug.
* The subject has evidence of acute intracranial or intratumoral hemorrhage either by MRI or computerized tomography (CT) scan. Subjects with resolving hemorrhage changes, punctate hemorrhage, or hemosiderin are eligible.
* The subject is unable to undergo MRI scan (eg, has pacemaker).
* The subject has received enzyme-inducing anti-epileptic agents within 14 days of study drug (eg, carbamazepine, phenytoin, phenobarbital, primidone).
* Patients whose only lesion undergoing resection has received stereotactic radiation within the past 3 months
* The subject has received any of the following prior anticancer therapy:

  * Biologic agents (antibodies, immune modulators, vaccines, cytokines) within 21 days prior to first dose of study drug
  * Prior treatment with Sacituzumab Govitecan
* Patients receiving UGT1A1 (Uridine diphosphate glucuronosyl transferase 1A1) inhibitors or inducers.
* History of significant cardiovascular disease, defined as:

  * Congestive heart failure greater than New York Heart Association (NYHA) Class II according to the NYHA Functional Classification.
  * Unstable angina or myocardial infarction within 6 months before enrollment.
  * Serious cardiac arrhythmia.
* Clinically significant ECG abnormality, including:

  * Marked Baseline prolonged QT/QTc interval (ie, a repeated demonstration of a QTc interval >500 ms) demonstrated on ECG at Screening.
  * History of risk factors for torsade de pointes (eg, heart failure, hypokalemia, family history of long QT Syndrome).
* Any medical or other condition which, in the opinion of the Investigator, causes the subject to be medically unfit to receive Sacituzumab Govitecan, or unsuitable for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Ratio of SN-38 and its metabolites relative to serum concentration | Day 1 of each 21 day cycle
  Levels of SN-38 and its metabolites will be measured and a ratio calculated relative to the serum concentration of SN-38 and its metabolites. The ratio will show the amount of investigational product that crosses the blood brain barrier to reach the tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Brenner, MD, PhD, Principal Investigator — University of Texas Health at San Antonio
Locations (1):
- Mays Cancer Center, UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Balinda HU, Kelly WJ, Kaklamani VG, Lathrop KI, Canola MM, Ghamasaee P, Sareddy GR, Michalek J, Gilbert AR, Surapaneni P, Tiziani S, Pandey R, Chiou J, Lodi A, Floyd JR 2nd, Brenner AJ. Sacituzumab Govitecan in patients with breast cancer brain metastases and recurrent glioblastoma: a phase 0 window-of-opportunity trial. Nat Commun. 2024 Aug 7;15(1):6707. doi: 10.1038/s41467-024-50558-9. PMID 39112464
- See also: Open Access publication of results — https://rdcu.be/dQe1F